CLINICAL TRIAL: NCT02353715
Title: PEAX: Men With Metastatic Castrate-Resistant Prostate Cancer Treated With Either Sipuleucel-T (Provenge®), Abiraterone Acetate (Zytiga®) or Enzalutamide (Xtandi®) Undergoing Cardiopulmonary EXercise Testing
Brief Title: Men With Metastatic Castrate-Resistant Prostate Cancer Treated With Either Sipuleucel-T (Provenge®), Abiraterone Acetate (Zytiga®) or Enzalutamide (Xtandi®) Undergoing Cardiopulmonary EXercise Testing
Acronym: PEAX
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00058229
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Abiraterone Acetate; sipuleucel-T

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Enzalutamide: Subjects will be administered enzalutamide per standard of care under the care of their treating physician. Cardiopulmonary Exercise Testing (CPET) will be performed at baseline and 21 weeks.
  Interventions: Drug: Enzalutamide
- Abiraterone: Subjects will be administered abiraterone acetate per standard of care under the care of their treating physician. Cardiopulmonary Exercise Testing (CPET) will be performed at baseline and 21 weeks.
  Interventions: Drug: Abiraterone acetate
- Sipuleucel-T: Subjects will be administered sipuleucel-T per standard of care under the care of their treating physician. Cardiopulmonary Exercise Testing (CPET) will be performed at baseline and 21 weeks.
  Interventions: Drug: Sipuleucel-T

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: Xtandi
  Groups: Enzalutamide
Drug: Abiraterone acetate
  Other Names: Zytiga
  Groups: Abiraterone
Drug: Sipuleucel-T
  Other Names: Provenge
  Groups: Sipuleucel-T

SUMMARY:
This is a pilot exercise physiology and quality of life study of subjects receiving standard of care therapy for their prostate cancer using FDA-approved drugs per their labeling (abiraterone, enzalutamide, or sipuleucel-T). Subjects with progressive, asymptomatic or minimally symptomatic mCRPC scheduled to be treated with either enzalutamide or abiraterone acetate for ≥3 months or a course of sipuleucel-T will be allocated to one of the treatments arms, according to the treatment chosen by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Male age ≥ 18 years
2. Histologically-confirmed adenocarcinoma of the prostate
3. Surgically or medically castrated
4. Starting either enzalutamide or abiraterone for at least 12 weeks OR starting a course of sipuleucel-T. Subjects being treated concomitantly with abiraterone or enzalutamide plus sipuleucel-T are eligible and should be enrolled on Arm A or Arm B, as appropriate.
5. ECOG performance status 0 or 1
6. Able to read and understand English, in the opinion of the treating provider, well enough to complete the study questionnaires
7. Able to comply with study requirements
8. Successful completion of a CPET in the opinion on the investigator

Exclusion Criteria:

1. Subjects who have had any surgical procedure (i.e. TURP, etc.) within 4 weeks prior to entering the study.
2. Subjects receiving treatment with BOTH abiraterone and enzalutamide
3. For Arm C (sipuleucel-T) only:

   1. subjects receiving abiraterone or enzalutamide concomitantly with sipuleucel-T should only be enrolled on Arm A or Arm B, as appropriate.
   2. subjects who have received prior sipuleucel-T
4. Subjects who are receiving any other investigational agents (i.e. enzalutamide or abiraterone plus an investigational drug).
5. Subjects with any of the following absolute contraindications to maximal exercise testing as recommended by the American Thoracic Society and the exercise testing guidelines for cancer subjects, in the opinion of the treating provider: (a) acute myocardial infarction (3-5 days), (b) unstable angina, (c) uncontrolled arrhythmias causing symptoms or hemodynamic compromise, (d) syncope, (e) acute endocarditis, (f) acute myocarditis or pericarditis, (g) uncontrolled heart failure, (h) acute pulmonary embolus or pulmonary infarction, (i) thrombosis of lower extremities, (j) suspected dissecting aneurysm, (k) uncontrolled asthma, (l) pulmonary edema, (m) room air desaturation at rest <85%, (n) respiratory failure, (o) acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise, (p) mental impairment leading to inability to cooperate, and (q) extensive bone metastases.
6. Significant cardiovascular disease, including:

   1. Symptomatic left ventricular dysfunction or known baseline left ventricular ejection fraction (LVEF) by multigated acquisition scan (MUGA) or echocardiogram (ECHO) of < lower limit of institutional normal (LLN). "Symptomatic" is defined as New York Heart Association (NYHA) Class II or greater. Note: MUGA and ECHCO do NOT need to be measured to establish eligibility for this study.
   2. Uncontrolled hypertension
   3. Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug
   4. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) within 12 months of first dose of study drug
   5. Uncontrolled cardiac arrhythmias
   6. Coronary or peripheral artery bypass graft within 6 months of first dose of study drug
   7. History of CVA, TIA, or rest claudication within 6 months of first dose of study drug
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
8. Known or suspected brain metastasis or leptomeningeal disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke clinics patients
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Change in VO2peak from baseline with abiraterone, enzalutamide or sipuleucel-T at week 21 | baseline, 21 weeks

SECONDARY OUTCOMES:
Compare VO2peak with patient- and physician reported functional status | 21 weeks
Evaluate the variability of CPET in all arms | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States